CLINICAL TRIAL: NCT06073925
Title: Use of Vitamin D as An Adjuvant Treatment in Children With Chronic Idiopathic Thrombocytopenic Purpura
Acronym: MansouraU
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MS.23.03.2332
Record Dates: First submitted 2023-05-14; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Immune Thrombocytopenia
Keywords: (ITP) Idiopathic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- chronic ITP children with VD level less than 30 ng/ml. (Active Comparator): will receive VD 3 50000 IU per week for 3 months beside their treatment for ITP.
  Interventions: Drug: VIT D
- chronic ITP children with VD level more than 30 ng/ml. (Active Comparator): will receive VD 3 50000 IU per week for 3 months beside their treatment for ITP.
  Interventions: Drug: VIT D
- Placebo (No Intervention): will receive their treatment for ITP.

INTERVENTIONS:
Drug: VIT D — 50000 IU per week of VIT D
  Other Names: Navigen
  Arms: chronic ITP children with VD level less than 30 ng/ml.; chronic ITP children with VD level more than 30 ng/ml.

SUMMARY:
Immune thrombocytopenia is an autoimmune disease in which platelets are targeted by the host immune system. Platelet depletion occurs when autoantibodies targeting glycoproteins (αIIb-β3 and GPIb) found on the surface of platelets opsonize the cells, resulting in destruction by macrophages. These antibodies can also bind to megakaryocytes and prevent complete maturation, which results in lowered levels of platelet production Vitamin D (VD) or 1,25-dihydroxyvitamin D, may be a potent immunomodulator, and it may have potential therapeutic use in many autoimmune diseases In 1991, researchers found that the production of interleukin (IL)-6 and IL-2 in cell cultures were reduced by 1,25(OH)2D3 VD deficiency is very common in children with either newly diagnosed or chronic ITP form.Correlation between hypovitaminosis D and a higher incidence of infections and autoimmune diseases was reported as well Case-Control interventional study (over time each participant will be randomized to be enrolled in one of either study arms in a random sequence). To evaluate the efficacy of VD supplementation as an adjuvant therapy in chronic ITP children and its effect on platelet count and bleeding score.

The participants will be - Children from 1 year to 18 years diagnosed with Chronic ITP with platelet count <100,000/microL.

Patients groups will be:

Patients of Chronic ITP aged from 1year till 18 years old . in this study will be divided into 2 groups ● Group A : All patients with VIT D insufficiency(The preferred level for 25(OH)D is now recommended by many experts to be >30 ng/ml) will receive supplementary Vitamin D3(NIVAGEN Vitamin D3 Cholecalciferol 50000 IU) oral once weekly for 3 months as adjuvant therapy in combination with their treatment for ITP.

● Group B : patients in this group have sufficient VIT D level and will be divided into 2 groups :

* Group 1 B :will receive their standard treatment for ITP with VIT D.
* Group 2 B :will receive their standard treatment for ITP without VIT D. Complete blood picture will be made at the beginning of study then monthly to evaluate the number of platelets that expected to increase after VD supplementation

DETAILED DESCRIPTION:
Introduction

Immune thrombocytopenia is an autoimmune disease in which platelets are targeted by the host immune system. Platelet depletion occurs when autoantibodies targeting glycoproteins (αIIb-β3 and GPIb) found on the surface of platelets opsonize the cells, resulting in destruction by macrophages. These antibodies can also bind to megakaryocytes and prevent complete maturation, which results in lowered levels of platelet production.

ITP of childhood is characterized by isolated thrombocytopenia (platelet count <100,000/microL with normal white blood cell count, hemoglobin, and blood smear).

The incidence of ITP in children is approximately 4-8 per 100,000 person-year . A recent history of viral illness is described in 50-65% of children with ITP. The peak age is 1-4 yr. ITP seems to occur more often in late winter and spring after the peak season of viral respiratory illness.

ITP can be classified by disease duration into; newly diagnosed (0-3 months), persistent (>3-12 months), or chronic (>12 months). The term "refractory" has been used to refer to patients who failed to improved after splenectomy.

Current treatment involves intravenous corticosteroids show efficacy in 50% to 80% of cases, but if treatment is stopped, the remission rate is only 10% to 30% immunosuppressants such as mycophenolate mofetil and azathioprine, cyclophosphamide, and intravenous immunoglobulin (IVIg).

Anti-D immunoglobulin that can only be given to RhD-positive individuals, thus limiting treatment options for RhD-negative persons. Rituximab has also been tried, and combinations of therapies have been used with some success .

If patients are refractory to drug treatments, splenectomy is a second line option; two-thirds of patients who undergo splenectomy for ITP respond to the treatment . However, complications may arise from this surgical procedure including hemorrhage, abscess, sepsis, thrombosis and death and relapse of ITP occurs in a median of 15% of patients .

Vitamin D (VD) or 1,25-dihydroxyvitamin D, may be a potent immunomodulator, and it may have potential therapeutic use in many autoimmune diseases . In 1991, researchers found that the production of interleukin (IL)-6 and IL-2 in cell cultures were reduced by 1,25(OH)2D3.

It was postulated that 1,25(OH) 2D3 may inhibit the production and function of IL-6 and, therefore, regulate lymphocyte functions. Activation of the vitamin D receptors (VDRs) is known to alter immune cell transcriptional patterns, proliferation and differentiation through several intracellular pathways . Both CD4+ and CD8+ lymphocytes contain significant amounts of VDRs, and thus it is reasonable to conclude that 1,25(OH)2D3 may play a role in the regulation of the immune response .

VD deficiency is very common in children with either newly diagnosed or chronic ITP form.Correlation between hypovitaminosis D and a higher incidence of infections and autoimmune diseases was reported as well.

There is an inverse association between TNF-α and VD levels in a healthy population and there is a protective association found for VD against inflammatory diseases such as inflamatory heart disease and rheumatoid arthritis. However, more studies are needed to precisely characterize the relationship between VD and TNF-α. Vitamin D therapy may show promise as adjunct to anti-TNF-α in autoimmune disease such as ITP .

Aim of the work:

To evaluate the efficacy of VD supplementation as an adjuvant therapy in chronic ITP children and its effect on platelet count and bleeding score.

Research gap:

To the best of our knowledge, no previous studies evaluating the effect of VD supplementation on chronic ITP children (only case reports).

Patients and methods

A randomized controlled trial will be conducted in the period from 2023 to 2024.

1. -Study design:

   Case-Control interventional study (over time each participant will be randomized to be enrolled in one of either study arms in a random sequence).
2. - Participants:

   A - Inclusion criteria:
   * Chirdren from 1 year to 18 years.
   * Diagnosed with Chronic ITP .
   * Platelet count <100,000/microL.

   B- Exclusion criteria:

   ● Other causes of thrombocytopenia.

   ● Acute and persistant ITP.

   ● Dysmorphic feature.

   ● Patients with other comorbidities.
3. -Study location:

Mansoura University Children Hospital- Hematology Out Patient Clinc. 4- Study duration:

Over one year from 2023 to 2024

5- Study methodology:

A- Randomization:

1. Procedure: Simple .
2. Allocation concealment: using sequentially numbered sealed envelop. 3- Sample size: pilot study.

B- Patients groups:

Patients of Chronic ITP aged from 1year till 18 years old . in this study will be divided into 2 groups ● Group A : All patients with VIT D insuffeciency(The preferred level for 25(OH)D is now recommended by many experts to be >30 ng/ml) will receive supplementary Vitamin D3(NIVAGEN Vitamin D3 Cholecalciferol 50000 IU) oral once weekly for 3 months as adjuvant therapy in combination with their treatment for ITP.

● Group B : patients in this group have suffecient VIT D level and will be divided into 2 groups :

* Group 1 B :will receive their standard treatment for ITP with VIT D.
* Group 2 B :will receive their standard treatment for ITP without VIT D.

Each patient in group A and group 1b will be provided with patient dairy to document patient's compliance:

1. Patients considered fulfilling >75% of the weekly oral VD their compliance will be considered (good compliance)
2. Patients fulfilling 50%-75% will be considered (fair compliance).
3. Patients fulfilling <50% will be considered (poor compliance).

C- History and examination:

1. Age.
2. Sex.
3. Duration of the illness.
4. Bleeding score, Each patient will be undergone examination for bleeding manifestation, bleeding score will be done for all patients and assessment of patients for growth parameters according to Table (1) Table (1): Scale of Bolton-Maggs and Moon -for severity of bleeding.

   None/mild ▪ No bleeding at all or bruising, petechiae, occasaional mild epistaxis with very little or no interference with daily living.

   Moderate ▪ More severe skin manifestation with some mucosal bleeding and more troublesome epistaxis or menorrhagia.

   Sever ▪ Bleeding episodes (epistaxis, melena, menorrhagia, and - or intracranial hemorrhage ) requiring hospital admission and - or blood transfusion, that is symptoms interfering seriously with quality of life.
5. Current treatment.
6. Examination for any bleeding signs.

D- laboratory assessment:

* Complete blood picture at the begining of study then monthly.
* Estimation of Vitamin D level by ELISA .

Ethical consideration:

Privacy was maintained by identification of the patients by coded numbers and all private data of the patients such as name, address and phone numbers didn't appear in the research instead, a code number was assigned to identify research participant.

The study protocol will be subjected for approval from Institutional Review Board of faculty of medicine - Mansoura University .

The merits of the study were explained to the participant.

The subjects that were involved in the research had the right to withdraw from the study at any time.

An informed consent obtained from all parents before enrollment of their children in the study.

Statistical Analysis :

All data will be collected, processed &analyzed using SPSS version 20. Quantitative data will be expressed as mean ±SD for parametric & median (minimum - maximum) for non-parametric, after testing norm- ality using Kolmogrov- Smirnov test. Categorical variables will be

described as number & percentage. The proper statistical test will be applied according to data. All tests will be 2 tailed & P value will be considered significant < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Chirdren from 1 year to 18 years.
* Diagnosed with Chronic ITP .
* Platelet count <100,000/microL.

Exclusion Criteria:

* Other causes of thrombocytopenia.
* Acute and persistant ITP.
* Dysmorphic feature.
* Patients with other comorbidities.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Participants who receive vitamin D will show change platelet count more than placepo group | 3 month
  To evaluate the efficacy of VD supplementation as an adjuvant therapy in chronic ITP children and its effect on platelet count and bleeding score.